CLINICAL TRIAL: NCT06605482
Title: Early Fixation for Diaphyseal Humeral Shaft Fractures in the Elderly Patients: A Prospective Cohort Study
Brief Title: Early Fixation for Diaphyseal Humeral Shaft Fractures in the Elderly Patients
Status: Recruiting | Type: Observational
Sponsor: Fraser Orthopaedic Research Society (Network)
Responsible Party: Sponsor
Other Study IDs: 2024137
Record Dates: First submitted 2024-09-11; First posted 2024-09-20 (Actual); Last update posted 2025-02-28 (Actual); Status verified 2025-02

CONDITIONS: Humerus Shaft Fracture; Elderly (People Aged 65 or More)
Keywords: patient outcomes
MeSH Terms: interventions — Patient Reported Outcome Measures; Range of Motion, Articular

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (2):
- Operative: Humeral shaft fracture is surgically managed with open reduction internal fixation or intramedullary nailing.
  Interventions: Other: Patient Reported Outcome Measures; Other: Range of Motion
- Non-operative: Humeral shaft fracture is conservatively managed with bracing or splinting
  Interventions: Other: Patient Reported Outcome Measures; Other: Range of Motion

INTERVENTIONS:
Other: Patient Reported Outcome Measures — Participants will complete the following outcome measures American Shoulder and Elbow Surgeons Evaluation Questionnaire - upper limb function score 12-Item Short Form Survey - general health questionnaire
Other: Range of Motion — Shoulder and Elbow Range of Motion collected at the time of radiographic union

SUMMARY:
The study purpose is to evaluate whether early surgical fixation of upper arm fractures in elderly patients' age 65 years and older improves patient functional and psychological outcome scores compared to the standard of care with non-operative management.

DETAILED DESCRIPTION:
A prospective cohort study following patients that are 65 years or older after they have suffered a humeral shaft fracture. Follow up will continue until 1 year post treatment to see functional and psychological outcomes.

ELIGIBILITY:
Inclusion Criteria:

1. Diaphyseal humeral shaft fracture (as defined as superior border of insertion of pectoralis major proximally, to the distal diaphysis)
2. Ambulatory (with or without the use of walking aides)

Exclusion Criteria:

1. Fractures with intra-articular extension
2. Ipsilateral upper extremity injury
3. Patients with vascular injury
4. Brachial plexus injury
5. Compartment syndrome
6. Pathological fractures
7. Open fractures
8. Periprosthetic fracture
9. BMI >40
10. Dementia or cognitive impairment that inhibits the collection of outcome measures
11. Likely problems, in the judgement of the investigator, with maintaining follow-up (i.e. patients with no fixed address, not mentally competent to give consent, intellectually challenged, patients without adequate support, etc.)
12. Inability to provide informed consent

Min Age: 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Study Population: Patients who present to the Royal Columbian Hospital or the investigators clinic with a diaphysial humeral shaft fracture.
Sampling Method: Probability Sample
Enrollment: 94 (Estimated)
Dates: Start 2024-11-07 (Actual); Primary Completion 2027-09-30 (Estimated); Study Completion 2027-12-31 (Estimated)

PRIMARY OUTCOMES:
American Shoulder and Elbow Score | Enrolment to 12 months post treatment
  Patient reported outcome measure for shoulder and elbow function. The score ranges from 0 to 100, with 0 the lowest level of function and 100 the highest level of function.

SECONDARY OUTCOMES:
12-Item Short Form Survey | Enrolment to 12 months post treatment
  General health patient reported outcome measure. Scores range from 0 to 100, with higher scores indicating better physical and mental health functioning.
Range of Motion | 3 months post treatment
  range of motion of shoulder and elbow

CONTACTS AND LOCATIONS:
Locations (1):
- Royal Columbian Hospital, New Westminster, British Columbia, Canada

IPD SHARING:
Plan to Share IPD: Undecided